CLINICAL TRIAL: NCT04217811
Title: Late Neutropenia in VLBW Preterm Babies - Characterization and Post Natal Menagement
Brief Title: Late Neutropenia in VLBW Preterm Babies
Status: Completed | Type: Observational
Sponsor: Hillel Yaffe Medical Center (Other Government)
Responsible Party: Principal Investigator, Erez Nadir, MD, Principal investigator, Hillel Yaffe Medical Center
Other Study IDs: 0160-19-HYMC
Record Dates: First submitted 2020-01-02; First posted 2020-01-03 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2021-08

CONDITIONS: Neutropenia
Keywords: VLBW; Neutropenia
MeSH Terms: conditions — Neutropenia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Late neutropenia: Neutrophil count < 1500
  Interventions: Other: No intervention
- No late neutropenia: Neutrophil count > 1500
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
There are rare reports regarding late neutropenua in very low birth weight preterm infants.

The investigators wish to characterize it among our population, and assess its consequenses and the postnatal menagement of the infants.

DETAILED DESCRIPTION:
There are rare reports regarding late neutropenua in very low birth weight preterm infants.

The investigators wish to characterize it among our population, and assess its consequenses and the postnatal menagement of the infants.

ELIGIBILITY:
Inclusion Criteria:

* Preterm infant with birth weight up to 1500 gram

Exclusion Criteria:

* Early neutroenia - neutrophil count < 1500 at the first week

Max Age: 30 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: VLBW infants
Sampling Method: Non-Probability Sample
Enrollment: 237 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Length of stay | 2 weeks
  Number of days

CONTACTS AND LOCATIONS:
Overall Officials: Erez Nadir, MD, Principal Investigator — Hillel Yaffe Medical Center
Locations (1):
- Hillel Yaffe medical center, Hadera, Hadera, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Juul SE, Calhoun DA, Christensen RD. "Idiopathic neutropenia" in very low birthweight infants. Acta Paediatr. 1998 Sep;87(9):963-8. doi: 10.1080/080352598750031635. PMID 9764892